CLINICAL TRIAL: NCT03439774
Title: Comparative Study of the Topcon Tonometers CT-800 and TRK-2P and the Haag-Streit Goldmann Manual Tonometer (Predicate) to Demonstrate Conformance to ANSI Z80.10-2014 Ophthalmic Instruments - Tonometers, to the FDA Guidance for Industry and FDA Staff, Tonometer-Premarket Notification [510(k)] Submissions, and to the Applicable Supplemental Information Sheet and Comparison of Pachymetry Values for Topcon TRK-2P With the Topcon SP-1P (Predicate)
Brief Title: Comparative Study of the Topcon Tonometers CT-800 and TRK-2P and the Haag-Streit Goldmann Manual Tonometer and Topcon SP-1P
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Topcon-TON-US-0002
Record Dates: First submitted 2017-12-08; First posted 2018-02-20 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Adults 18 years old or older
  Interventions: Device: Topcon CT-800; Device: Topcon TRK-2P

INTERVENTIONS:
Device: Topcon CT-800 — tonometer
Device: Topcon TRK-2P — tonometer, pachymeter

SUMMARY:
The study will assess the CT-800 and TRK-2P for conformity to ANSI Z80.10-2014 Ophthalmic Instruments - Tonometers, to the FDA Guidance for Industry and FDA Staff, Tonometer-Premarket Notification [510(k)] Submissions, and to the applicable Supplemental Information Sheet. This clinical device study will also assess the substantial equivalence of TRK-2P to a predicate device in regard to pachymetry.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years of age of either sex and any race or ethnicity;
2. be willing and able to provide written informed consent prior to any study procedures being performed;
3. be willing and able to follow all instructions and attend all study visits;

Exclusion Criteria:

1. have only one functional eye;
2. have poor or eccentric fixation in either eye;
3. have corneal scarring or have had corneal surgery, including corneal laser surgery in either eye;
4. have microphthalmos in either eye;
5. have buphthalmos in either eye;
6. be a contact lens wearer, meaning having worn soft contact lenses within the past 3 months and/or rigid permeable gas lenses within the past 6 months;
7. have dry eyes, meaning having been diagnosed by a physician with dry eyes and currently using a prescribed medication or daily use of an artificial tear;
8. be a lid squeezer - blepharospasm;
9. have nystagmus in either eye;
10. have keratoconus in either eye;
11. have any other corneal or conjunctival pathology or infection in either eye;
12. have a condition or a situation, which in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 250 subjects will have both of their eyes measured.
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Agreement of IOP | 1 day
  Agreement of the measured IOP between the test devices and the predicate device for the tonometer function of CT-800 and TRK-2P. Presentation of results and analyses will include descriptive statistics (mean, standard deviation, limits of agreement), Bland-Altman plot and linear regression.
Agreement of Corneal Thickness | 1 day
  Agreement of measured corneal thickness between the test device and the predicate device for the pachymeter function of the TRK-2P. Presentation of results and analyses will include descriptive statistics (mean, standard deviation, limits of agreement), Bland-Altman plot and Deming regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States